CLINICAL TRIAL: NCT05837858
Title: Study on Biomarkers of Whole Grain Dietary Intake in Chinese Population
Brief Title: The Human Metabolic Profile and Gut Microbiota Under Various Dietary Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: xuyajun197673
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-04

CONDITIONS: Biomarkers
Keywords: Food biomarker; Whole grain; Chinese population

STUDY DESIGN:
Intervention Model Description: Randomized Crossover Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole grain-wheat flour food, then refined wheat flour food (Experimental): Participants first received food made by 50 g whole grain wheat flour during breakfast in a fasting state. Standardized meals were provided to the volunteers from the dinner of the day before the intervention day, as well as up to 48 h after the administration of the test food. After a washout period of 5 days, volunteers followed a 2-day restricted diet before the intervention day. Participants then received food made by 50 g refined grain wheat flour in a fasting state.
  Interventions: Other: whole grain-wheat flour food+standardized meals; Other: refined wheat flour food+standardized meals
- refined wheat flour food, then whole grain-wheat flour food (Experimental): Participants first received food made by 50 g refined grain wheat flour during breakfast in a fasting state. Standardized meals were provided to the volunteers from the dinner of the day before the intervention day, as well as up to 48 h after the administration of the test food. After a washout period of 5 days, volunteers followed a 2-day restricted diet before the intervention day. Participants then received food made by 50 g whole grain wheat flour in a fasting state.
  Interventions: Other: whole grain-wheat flour food+standardized meals; Other: refined wheat flour food+standardized meals

INTERVENTIONS:
Other: whole grain-wheat flour food+standardized meals — whole grain food made by 50 g whole grain wheat flour
Other: refined wheat flour food+standardized meals — refined grain food made by 50 g refined wheat flour

SUMMARY:
The goal of this food intervention study is to screen/validate the whole grain food intake biomarker in health Chinese's population.

DETAILED DESCRIPTION:
Although increased consumption of whole grains (WGs) is associated with improved health outcomes, the dietary intake assessment and health mechanisms for WGs or WG-containing food remain unresolved. In addition, information regarding its consumption and health effects in Chinese people is scarce. Biomarkers of WGs intake would allow a more accurate assessment of its consumption in nutrition studies. The investigators want to perform a crossover study where participants were subjected to a WG-wheat flour or a refine wheat-flour Chinese diet. Using a metabolomics approach, the investigators aimed to identify the WG-specific metabolites present in plasma/urine after consumption WG or WG foods, including new candidate biomarkers of WG intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* age 18-40 years
* BMI 18.5-23.9 kg/m2.

Exclusion Criteria:

* pregnancy or breastfeeding
* vegetarian;
* smokers;
* acute and chronic diseases;
* allergic to wheat;
* frequent nutrients supplement use;
* medication use of antibiotics within 1-month;
* more than 3 kg weight change within 3-month;
* unwillingness to follow dietary restrictions;

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Changes in metabolite profiles present in blood plasma and urine before the dietary intervention and in kinetics over 24 hours. | Baseline and 0-24 hours after intervention food intake
  Metabolite profiles analyzed using a non-targeted metabolomics approach and targeted metabolomics approach with a Orbitrap Mass Analyzer. Blood plasma samples collected at time 0 hours, 2 hours, 4 hours, and 24 hours. Urine fractions collected at 0-2 hours, 2-4 hours, 4-6 hours, 6-9 hours, 9-12 hours, 12-24 hours and 24-48 hours. Identification of biomarkers of acute intake of the foods of interest through the comparison of specific metabolomes after single dose of WG food or refined grain food in Chinese population.

SECONDARY OUTCOMES:
The influence of gut flora on whole grain markers | after the administration of the test meal
  Gut flora abundance and metabolites level correlation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yunjia yang, Principal Investigator — Peking University; Yalin Zhou, Principal Investigator — Peking University
Locations (1):
- Department of Nutrition and Food Hygiene, School of Public Health, Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Shared IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: December 30, 2023
Access Criteria: In a publication